CLINICAL TRIAL: NCT02457065
Title: Skin Care Behaviors Among Melanoma Survivors and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Michael S. Chapman, Staff Physician, Dermatology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00028495 D15090
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Melanoma
Keywords: survivors; family
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive Plaque (Experimental): Treatment
  "Melanoma Survivor" plaque: After the patients enrolled in the study and completed the initial survey, the investigators gave the patients a small 3.5 by 2 inch wooden plaque that celebrates their survival of melanoma and reminds them to engage in skin cancer prevention behaviors.
  Interventions: Behavioral: "Melanoma Survivor" plaque
- Do Not Receive Plaque (No Intervention): Control
  No "Melanoma Survivor" plaque: After the patients enrolled in the study and completed the initial survey, the investigators did not give the patients a small 3.5 by 2 inch wooden plaque that celebrates their survival of melanoma and reminds them to engage in skin cancer prevention behaviors or any other intervention.

INTERVENTIONS:
Behavioral: "Melanoma Survivor" plaque — The investigators give the patients a small 3.5 by 2 inch wooden plaque that celebrates their survival of melanoma and reminds them to engage in skin cancer prevention behaviors.
  Other Names: Receive Plaque
  Arms: Receive Plaque

SUMMARY:
A patient's sun-related behavior greatly influences the likelihood of that patient developing melanoma, the most dangerous form of skin cancer. Prior research shows current educational strategies on inducing preventative behaviors such as wearing sun-protection clothing and wearing sunscreen are inadequate at effectively changing behavior when used in isolation -- patients are aware of the dangers of not engaging in these preventative measures but forgo them nonetheless.

The investigators are researching methods to positively influence skin cancer prevention behaviors among melanoma survivors and their families. The first objective of this study is to compare patient and familial sun exposure and cancer screening activity before and after a patient's diagnosis with primary melanoma. The second objective of this study is to note if hanging a "Melanoma Survivor" plaque in a melanoma survivor's bathroom will significantly affect the survivor's and broader family's sun exposure and cancer screening activity.

The investigators' sample of patients consists of survivors of primary cutaneous melanoma less than 4.0 mm in depth who came through the Dermatology Clinic at Dartmouth-Hitchcock Medical Center and voluntarily chose to participate in the study after being informed of the nature of the research. These patients completed a confidential survey assessing sun exposure related activities immediately before and after their diagnosis. After the participants filled out the survey, the investigators asked the participants if they could nominate a family member to whom the investigators could explain the purpose of this research study to and confidentially ask an additional set of questions to evaluate the broader impact of a melanoma diagnosis. From the investigators' original sample, the investigators randomly chose a few families who would display the survivor plaque in their primary bathroom. After six-to-twelve months, during the each patient's follow up visit, the investigators asked the patient and the patient's nominated family member to fill out another survey to assess sun exposure related activity.

On the surveys, no names were recorded. Everything was anonymous.

DETAILED DESCRIPTION:
This study is investigating a method to positively influence skin cancer prevention behaviors among melanoma survivors and their families. The first objective is to compare patient and familial sun exposure and cancer screening activity before and after a patient's diagnosis with primary cutaneous melanoma less than 4.0 mm in depth. It is believed that the diagnosis will positively affect behavior regarding skin cancer prevention as the diagnosis of melanoma makes the risk associated with sun-exposure and skin cancer a tangible issue. The second objective is to test whether receiving a "Melanoma Survivor" plaque and posting it in a melanoma survivor's bathroom will significantly affect the survivor's and broader family's sun exposure and cancer screening activity. Marketing research has shown similar techniques have been effective in causing individuals to consume goods (e.g. getting free pens with company logos makes you more likely to buy goods from that company), and the investigators think such techniques are transferable into the field of public health.

ELIGIBILITY:
Inclusion Criteria:

* patient has melanoma diagnosis within past 10 years less than 4mm in depth

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Chapman, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center (Heater Road), Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Survivors of primary cutaneous melanoma less than 4.0 mm in depth who came through the Dermatology Clinic at Dartmouth-Hitchcock Medical Center and voluntarily chose to participate in the study after being informed of the nature of the research.
Pre-assignment Details: All enrolled participants were assigned to arms/groups. None were excluded from the study.
Groups:
- Receive Plaque: Treatment
  After the patients enrolled in the study and completed the initial survey, the investigators gave the patients a small 3.5 by 2 inch wooden plaque that celebrates their survival of melanoma and reminds them to engage in skin cancer prevention behaviors.
- Do Not Receive Plaque: Control
  After the patients enrolled in the study and completed the initial survey, the investigators did not give the patients a small 3.5 by 2 inch wooden plaque that celebrates their survival of melanoma and reminds them to engage in skin cancer prevention behaviors or any other intervention.
Period: Overall Study
Arm/Group | Receive Plaque | Do Not Receive Plaque
Started | 27 | 27
Completed | 18 | 16
Not Completed | 9 | 11
Not completed — Lost to Follow-up | 9 | 11

BASELINE CHARACTERISTICS:
Population: Survivors of primary cutaneous melanoma less than 4.0 mm in depth who came through the Dermatology Clinic at Dartmouth-Hitchcock Medical Center and voluntarily chose to participate in the study after being informed of the nature of the research.
Groups:
- Total: Total of all reporting groups
Arm/Group | Receive Plaque | Do Not Receive Plaque | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Customized [Count of Participants; unit: Participants] — Population: Age was not collected from any participant.
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Sex/Gender were not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Influence of a Patient's Melanoma Diagnosis on the Survivor's and Broader Family's Skin Cancer Prevention Activity.
Description: Subjects filled out a survey when they enrolled in the study assessing their skin cancer prevention behaviors. Survey questions asked the patient and a family member of theirs to comment on patient and familial sun exposure and cancer screening activity before and after the patient's diagnosis with primary melanoma. Subjects self-reported if the diagnosis changed their behavior.
Time Frame: Collected via a survey administered immediately after a subject enrolled in the study.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Receive Plaque | Do Not Receive Plaque
Number analyzed (Participants) | 27 | 27
Participants
  Diagnosis changed patient prevention behavior: Yes | 24 | 22
  Diagnosis changed patient prevention behavior: No | 2 | 5
  Diagnosis changed patient prevention behavior: Unsure | 1 | 0
  Diagnosis changed familial prevention behavior: Yes | 18 | 15
  Diagnosis changed familial prevention behavior: No | 6 | 9
  Diagnosis changed familial prevention behavior: Unsure | 3 | 3

2. Primary Outcome: Influence of a "Melanoma Survivor" Plaque on the Survivor's and Broader Family's Skin Cancer Prevention Activity.
Description: Subjects filled out a survey when they enrolled in the study assessing their skin cancer prevention behaviors. The investigators randomly gave some subjects a "Melanoma Survivor" plaque. After 6-12 months, the subjects again filled out a survey assessing their skin cancer prevention behaviors. The investigators analyzed the difference in each subject's responses to the same survey questions over time. The investigators then analyzed the difference between the responses of the subjects who saw the plaque and the subjects who did not see the plaque to discern the influence of the plaque on skin cancer prevention behaviors. Survey questions asked the patient and a family member of theirs to comment on patient and familial sun exposure and cancer screening activity. Subjects self-reported if the their behavior changed over time.
Time Frame: 6-12 months between time of completion of first survey and second survey.
Population: Survivors of primary cutaneous melanoma less than 4.0 mm in depth who came through the Dermatology Clinic at Dartmouth-Hitchcock Medical Center, voluntarily chose to participate in the study after being informed of the nature of the research, and then completed the follow up survey 6-12 months after their initial enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Receive Plaque | Do Not Receive Plaque
Number analyzed (Participants) | 18 | 16
Participants
  Patient prevention behavior changed over time: Yes | 9 | 4
  Patient prevention behavior changed over time: No | 7 | 11
  Patient prevention behavior changed over time: Unsure | 2 | 1
  Familial prevention behavior changed over time: Yes | 8 | 4
  Familial prevention behavior changed over time: No | 8 | 10
  Familial prevention behavior changed over time: Unsure | 2 | 2

ADVERSE EVENTS:
Time Frame: After six-to-twelve months, during the each patient's follow up visit at the Dermatology clinic.
Description: The researchers did not anticipate any risks to study participants other than those regularly encountered in day-to-day life. During the follow up survey, no participants stated that the study adversely affected them.
Groups:
- Receive Plaque: Treatment
  Sun protection behaviors: The investigators give the patients a small 3.5 by 2 inch wooden plaque that celebrates their survival of melanoma and reminds them to engage in skin-protective behaviors
- Do Not Receive Plaque: Control
  These patients did not receive any intervention from the investigators.
Arm/Group | Receive Plaque | Do Not Receive Plaque
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

LIMITATIONS AND CAVEATS:
Did not reach anticipated sample size due to difficulties related to enrollment and patient/family-member follow up, which led to the small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No